CLINICAL TRIAL: NCT01845649
Title: A Randomized, Multicenter, Double-Blind, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of WC3011 in Postmenopausal Women With Dyspareunia
Brief Title: Study to Evaluate Safety and Efficacy of WC3011 (Estradiol Vaginal Cream) in Postmenopausal Women With Dyspareunia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR-08112
Record Dates: First submitted 2013-04-25; First posted 2013-05-03 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2021-09

CONDITIONS: Vulvovaginal Atrophy
Keywords: Vulvovaginal Atrophy; Dyspareunia; Postmenopausal
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle (3 Times/Week) (Active Comparator): Vehicle applied to the vagina daily for 14 days followed by dosing 3 times per week for 10 weeks.
  Interventions: Drug: Vehicle
- WC3011 Estradiol Vaginal Cream (3 Times/Week) (Experimental): WC3011 Estradiol vaginal cream applied daily for 14 days followed by dosing 3 times per week for 10 weeks.
  Interventions: Drug: WC3011 Estradiol Vaginal Cream

INTERVENTIONS:
Drug: WC3011 Estradiol Vaginal Cream — Daily for 14 days followed by 3 times per week for 10 weeks
  Other Names: WC3011
  Arms: WC3011 Estradiol Vaginal Cream (3 Times/Week)
Drug: Vehicle — Daily for 14 days followed by 3 times per week for 10 weeks
  Arms: Vehicle (3 Times/Week)

SUMMARY:
The purpose of the study is to determine if WC3011 is safe and effective in treating the symptom of painful intercourse secondary to vulvovaginal atrophy as measured by participant self-assessment when compared to vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active with self-identified dyspareunia (pain with sexual activity), at least moderate to severe and most bothersome symptom of vulvovaginal atrophy (VVA)
* Postmenopausal and meets 1 of the following: 12 months spontaneous amenorrhea, 6 months spontaneous amenorrhea with FSH (follicle stimulating hormone) >40 mIU/mL,6 weeks postsurgical bilateral oophorectomy with confirmation by FSH >40 mIU/mL, surgical report or ultrasound, 6 weeks postsurgical hysterectomy with ovary failure confirmed by FSH >40 mIU/mL
* Age ≥40 years; ≥35 with bilateral oophorectomy
* Vaginal pH >5.0
* Less than or equal to 5% superficial cells on vaginal wall cytologic smear
* Normal clinical breast exam or negative mammogram if ≥ 40 years of age
* Negative urine pregnancy test (non-hysterectomized and <12 months amenorrhea)

Exclusion Criteria:

* Enrollment in Sponsor's Study PR-04409 or PR-05812
* Participation in clinical trial or use of investigational drug within 30 days prior to screening
* Known hypersensitivity to estrogen and/or progestin therapy
* Known or suspected premalignant or malignant disease or history steroid-dependent malignancy
* Manifestation or treatment for significant cardiovascular disease (congestive heart failure, stroke or ischemic attack, myocardial infarction, coronary artery bypass, percutaneous angioplasty or >50% angiographic narrowing of coronary artery
* Thrombophlebitis or thromboembolic disorder or history of
* Insulin-dependent diabetes mellitus
* Increased frequency or severity of headaches while on hormone or estrogen therapy
* Currently taking St. John's Wort
* Drug/alcohol addiction within past 2 years
* Treatment with anticoagulants (heparin or warfarin)
* Smoking ≥15 cigarettes/day

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2013-04-12 (Actual); Primary Completion 2013-11-20 (Actual); Study Completion 2013-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, PharmD, Study Director — Warner Chilcott
Locations (51):
- United States (51):
  - Warner Chilcott Investigational Study Site, Birmingham, Alabama
  - Warner Chilcott Investigational Study Site, Mobile, Alabama
  - Warner Chilcott Investigational Study Site, Chandler, Arizona
  - Warner Chilcott Investigational Study Site, Phoenix, Arizona
  - Warner Chilcott Investigational Study Site, Scottsdale, Arizona
  - Warner Chilcott Investigational Study Site, Tucson, Arizona
  - Warner Chilcott Investigational Study Site, Sacramento, California
  - Warner Chilcott Investigational Study Site, San Diego, California
  - Warner Chilcott Investigational Study Site, New London, Connecticut
  - Warner Chilcott Investigational Study Site, Washington D.C., District of Columbia
  - Warner Chilcott Investigational Study Site, Boynton Beach, Florida
  - Warner Chilcott Investigational Study Site, Clearwater, Florida
  - Warner Chilcott Investigational Study Site, Jacksonville, Florida
  - Warner Chilcott Investigational Study Site, Miami, Florida
  - Warner Chilcott Investigational Study Site, Ormond Beach, Florida
  - Warner Chilcott Investigational Study Site, Palm Beach Gardens, Florida
  - Warner Chilcott Investigational Study Site, Pinellas Park, Florida
  - Warner Chilcott Investigational Study Site, West Palm Beach, Florida
  - Warner Chilcott Investigational Study Site, Atlanta, Georgia
  - Warner Chilcott Investigational Study Site, Roswell, Georgia
  - Warner Chilcott Investigational Study Site, Savannah, Georgia
  - Warner Chilcott Investigational Study Site, Granger, Indiana
  - Warner Chilcott Investigational Study Site, Lexington, Kentucky
  - Warner Chilcott Investigational Study Site, Marrero, Louisiana
  - Warner Chilcott Investigational Study Site, New Orleans, Louisiana
  - Warner Chilcott Investigational Study Site, Kalamazoo, Michigan
  - Warner Chilcott Investigational Study Site, Chaska, Minnesota
  - Warner Chilcott Investigational Study Site, Las Vegas, Nevada
  - Warner Chilcott Investigational Study Site, Moorestown, New Jersey
  - Warner Chilcott Investigational Study Site, Greensboro, North Carolina
  - Warner Chilcott Investigational Study Site, New Bern, North Carolina
  - Warner Chilcott Investigational Study Site, Raleigh, North Carolina
  - Warner Chilcott Investigational Study Site, Winston-Salem, North Carolina
  - Warner Chilcott Investigational Study Site, Cincinnati, Ohio
  - Warner Chilcott Investigational Study Site, Cleveland, Ohio
  - Warner Chilcott Investigational Study Site, Columbus, Ohio
  - Warner Chilcott Investigational Study Site, Jenkintown, Pennsylvania
  - Warner Chilcott Investigational Study Site, Philadelphia, Pennsylvania
  - Warner Chilcott Investigational Study Site, Pittsburgh, Pennsylvania
  - Warner Chilcott Investigational Study Site, Warwick, Rhode Island
  - Warner Chilcott Investigational Study Site, Bluffton, South Carolina
  - Warner Chilcott Investigational Study Site, Greer, South Carolina
  - Warner Chilcott Investigational Study Site, Austin, Texas
  - Warner Chilcott Investigational Study Site, Dallas, Texas
  - Warner Chilcott Investigational Study Site, Houston, Texas
  - Warner Chilcott Investigational Study Site, San Antonio, Texas
  - Warner Chilcott Investigational Study Site, South Jordan, Utah
  - Warner Chilcott Investigational Study Site, Norfolk, Virginia
  - Warner Chilcott Investigational Study Site, Richmond, Virginia
  - Warner Chilcott Investigational Study Site, Seattle, Washington
  - Warner Chilcott Investigational Study Site, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
Started | 273 | 277
Safety Population | 271 | 277
Modified Intent-to-treat (mITT) Population | 233 | 239
Completed | 242 | 255
Not Completed | 31 | 22
Not completed — Adverse Event | 7 | 10
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrew Consent | 12 | 4
Not completed — Protocol Deviation | 7 | 4
Not completed — Reason not Specified | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included participants who were randomized into the study and took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week) | Total
Number analyzed (Participants) | 271 | 277 | 548
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (6.1) | 58.7 (6.4) | 58.6 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 271 | 277 | 548
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Participant's Self-Assessment of Symptom of Vulvovaginal Atrophy (VVA): Dyspareunia (Pain Associated With Sexual Activity) to Final Assessment
Description: Participant's self-assessment of the symptom of VVA (dyspareunia) was scored on a 4-point scale where: 0=none, 1=mild, 2=moderate or 3=severe. Higher score indicates the most bothersome symptoms. A negative change from Baseline indicates improvement. Final Assessment is defined as the last available post-baseline assessment for the given efficacy endpoint.
Time Frame: Baseline (Day 0) to final assessment (Up to Week 12)
Population: Modified Intent-to-treat (mITT) Population included participants in the Safety population who had at least 1 postbaseline primary efficacy assessment and met all of the following inclusion criteria: ≤5% superficial cells on a vaginal wall smear, a vaginal pH >5.0, and the participants most bothersome symptom of VVA was dyspareunia with moderate to severe intensity. Number analyzed is the number of participants with available data at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
Number analyzed (Participants) | 233 | 239
score on a scale
  Baseline | 2.7 (0.44) | 2.7 (0.45)
  Change from Baseline to Final Assessment: number analyzed (Participants) | 229 | 231
  Change from Baseline to Final Assessment | -1.2 (0.93) | -1.5 (0.97)

2. Primary Outcome: Change From Baseline in Vaginal pH to Final Assessment
Description: Vaginal pH was obtained at baseline and final visit of the study. The pH was a numeric value from 0 to 14 expressing the acidity or alkalinity of the vaginal fluids where 7 was neutral, lower values were more acidic (values of 0-6) and higher values more alkaline (values of 8-14). A negative change from Baseline indicates improvement. Final Assessment is defined as the last available post-baseline assessment for the given efficacy endpoint.
Time Frame: Baseline (Day 0) to final assessment (Up to Week 12)
Population: mITT Population included participants in the Safety population who had at least 1 postbaseline primary efficacy assessment and met all of the following inclusion criteria: ≤5% superficial cells on a vaginal wall smear, a vaginal pH >5.0, and the participants most bothersome symptom of VVA was dyspareunia with moderate to severe intensity. Number analyzed is the number of participants with available data at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
Number analyzed (Participants) | 233 | 239
score on a scale
  Baseline | 6.35 (0.66) | 6.37 (0.66)
  Change from Baseline to Final Assessment: number analyzed (Participants) | 225 | 232
  Change from Baseline to Final Assessment | -0.53 (0.92) | -1.36 (0.89)

3. Primary Outcome: Change From Baseline in the Percentage of Vaginal Superficial Cells to Final Assessment
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of superficial cells. A positive change from Baseline indicates improvement. Final assessment is defined as the last available postbaseline assessment.
Time Frame: Baseline (Day 0) to final assessment (Up to Week 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
Number analyzed (Participants) | 233 | 239
percentage of superficial cells
  Baseline | 0.2 (0.75) | 0.2 (0.70)
  Change from Baseline to Final Assessment: number analyzed (Participants) | 221 | 217
  Change from Baseline to Final Assessment | 1.4 (6.08) | 10.1 (16.72)

4. Primary Outcome: Change From Baseline in the Percentage of Vaginal Parabasal Cells to Final Assessment
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of parabasal cells. A negative change from Baseline indicates improvement. Final assessment is defined as the last available postbaseline assessment.
Time Frame: Baseline (Day 0) to final assessment (Up to Week 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
Number analyzed (Participants) | 233 | 239
percentage of parabasal cells
  Baseline | 50.6 (43.09) | 53.5 (42.00)
  Change From Baseline to Final Assessment: number analyzed (Participants) | 221 | 217
  Change From Baseline to Final Assessment | -14.6 (39.55) | -48.5 (45.11)

5. Secondary Outcome: Change From Baseline in Participant's Self-Assessment of the Symptom of VVA: Dyspareunia to Weeks 2, 4, 8, and 12
Description: Participant's self-assessment of the symptom of VVA (dyspareunia) was scored on a 4-point scale where: 0=none, 1=mild, 2=moderate or 3=severe. Higher score indicates the most bothersome symptoms. A negative change from Baseline indicates improvement.
Time Frame: Baseline to Weeks 2, 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
Number analyzed (Participants) | 233 | 239
score on a scale
  Baseline | 2.7 (0.44) | 2.7 (0.45)
  Change From Baseline to Week 2: number analyzed (Participants) | 201 | 207
  Change From Baseline to Week 2 | -0.8 (0.87) | -0.8 (0.89)
  Change From Baseline to Week 4: number analyzed (Participants) | 203 | 208
  Change From Baseline to Week 4 | -1.1 (0.93) | -1.2 (0.93)
  Change From Baseline to Week 8: number analyzed (Participants) | 204 | 209
  Change From Baseline to Week 8 | -1.2 (0.92) | -1.5 (0.96)
  Change From Baseline to Week 12: number analyzed (Participants) | 200 | 201
  Change From Baseline to Week 12 | -1.2 (0.90) | -1.5 (0.95)

6. Secondary Outcome: Change From Baseline in Participant's Self-Assessment of the Other Symptoms of VVA to Weeks 2, 4, 8, 12, and Final Assessment
Description: Self-Assessment of the symptoms of VVA, other than dyspareunia and vaginal bleeding associated with sexual activity, (vaginal and/or vulvar irritation/itching, dysuria and vaginal dryness) were evaluated by a questionnaire. Each symptom was scored on a 4-point scale where: 0=none, 1=mild, 2=moderate or 3=severe. Higher scores indicate the most bothersome symptoms. A negative change from Baseline indicates improvement. Final Assessment is defined as the last available post-baseline assessment for the given efficacy endpoint.
Time Frame: Baseline (Day 0) to Weeks 2, 4, 8, 12, and final assessment (Up to Week 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
Number analyzed (Participants) | 233 | 239
score on a scale
  Vaginal Itching-Baseline | 0.9 (0.89) | 1.0 (0.89)
  Vaginal Itching-Change From Baseline to Week 2: number analyzed (Participants) | 229 | 238
  Vaginal Itching-Change From Baseline to Week 2 | -0.3 (0.94) | -0.3 (0.94)
  Vaginal Itching-Change From Baseline to Week 4: number analyzed (Participants) | 225 | 236
  Vaginal Itching-Change From Baseline to Week 4 | -0.5 (0.94) | -0.3 (0.96)
  Vaginal Itching-Change From Baseline to Week 8: number analyzed (Participants) | 220 | 228
  Vaginal Itching-Change From Baseline to Week 8 | -0.5 (0.98) | -0.4 (0.97)
  Vaginal Itching-Change From Baseline to Week 12: number analyzed (Participants) | 214 | 219
  Vaginal Itching-Change From Baseline to Week 12 | -0.6 (0.95) | -0.4 (0.96)
  Vaginal Itching-Change From Baseline to Final Assessment: number analyzed (Participants) | 232 | 239
  Vaginal Itching-Change From Baseline to Final Assessment | -0.5 (0.98) | -0.4 (0.95)
  Dysuria-Baseline | 0.4 (0.74) | 0.4 (0.72)
  Dysuria-Change From Baseline to Week 2: number analyzed (Participants) | 229 | 238
  Dysuria-Change From Baseline to Week 2 | -0.1 (0.82) | -0.1 (0.77)
  Dysuria-Change From Baseline to Week 4: number analyzed (Participants) | 225 | 236
  Dysuria-Change From Baseline to Week 4 | -0.2 (0.76) | -0.1 (0.80)
  Dysuria-Change From Baseline to Week 8: number analyzed (Participants) | 220 | 228
  Dysuria-Change From Baseline to Week 8 | -0.2 (0.73) | -0.2 (0.76)
  Dysuria-Change From Baseline to Week 12: number analyzed (Participants) | 214 | 219
  Dysuria-Change From Baseline to Week 12 | -0.2 (0.78) | -0.2 (0.75)
  Dysuria-Change From Baseline to Final Assessment: number analyzed (Participants) | 232 | 239
  Dysuria-Change From Baseline to Final Assessment | -0.2 (0.80) | -0.2 (0.72)
  Vaginal Dryness-Baseline | 2.3 (0.80) | 2.3 (0.73)
  Vaginal Dryness-Change From Baseline to Week 2: number analyzed (Participants) | 229 | 238
  Vaginal Dryness-Change From Baseline to Week 2 | -0.6 (1.08) | -0.7 (1.00)
  Vaginal Dryness-Change From Baseline to Week 4: number analyzed (Participants) | 225 | 236
  Vaginal Dryness-Change From Baseline to Week 4 | -0.8 (0.96) | -0.9 (0.91)
  Vaginal Dryness-Change From Baseline to Week 8: number analyzed (Participants) | 220 | 228
  Vaginal Dryness-Change From Baseline to Week 8 | -0.9 (0.98) | -1.1 (0.91)
  Vaginal Dryness-Change From Baseline to Week 12: number analyzed (Participants) | 214 | 219
  Vaginal Dryness-Change From Baseline to Week 12 | -0.9 (0.98) | -1.2 (0.94)
  Vaginal Dryness-Change From Baseline to Final Assessment | -0.8 (0.98) | -1.2 (0.97)

7. Secondary Outcome: Percentage of Participants With Vaginal Bleeding Associated With Sexual Activity at Each Visit
Description: Vaginal bleeding associated with sexual activity was assessed by participants as either "present" or "absent". Number of participants with assessment "present" are reported. Final Assessment is defined as the last available post-baseline assessment for the given efficacy endpoint.
Time Frame: Baseline (Day 0), Weeks 2, 4, 8, 12 and final assessment (Up to Week 12)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
Number analyzed (Participants) | 233 | 239
percentage of participants
  Baseline | 27.0 | 28.0
  Week 2: number analyzed (Participants) | 201 | 207
  Week 2 | 15.9 | 16.4
  Week 4: number analyzed (Participants) | 203 | 208
  Week 4 | 7.9 | 7.2
  Week 8: number analyzed (Participants) | 204 | 209
  Week 8 | 10.8 | 6.7
  Week 12: number analyzed (Participants) | 199 | 201
  Week 12 | 12.1 | 7.5
  Final Assessment: number analyzed (Participants) | 229 | 231
  Final Assessment | 14.4 | 6.5

8. Secondary Outcome: Change From Baseline in the Investigator's Assessment of Each of the Signs of VVA to Week 12 and Final Assessment
Description: Investigator's assessment of vaginal health was performed by visual inspection of the vagina with respect to the signs of VVA: atrophy, pallor, vaginal dryness, friability, and petechiae each graded on a 4-point scale where: 0=none, 1=mild, 2=moderate or 3=severe. Higher scores are worse. A negative change from Baseline indicates improvement. Final assessment is defined as the last available postbaseline assessment.
Time Frame: Baseline (Day 0) to Week 12 and Final assessment (Up to Week 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
Number analyzed (Participants) | 233 | 239
score on a scale
  Atrophy-Baseline: number analyzed (Participants) | 232 | 239
  Atrophy-Baseline | 2.0 (0.60) | 2.0 (0.64)
  Atrophy-Change From Baseline to Week 12: number analyzed (Participants) | 211 | 217
  Atrophy-Change From Baseline to Week 12 | -0.5 (0.75) | -0.9 (0.84)
  Atrophy-Change From Baseline to Final Assessment: number analyzed (Participants) | 226 | 233
  Atrophy-Change From Baseline to Final Assessment | -0.5 (0.75) | -0.9 (0.83)
  Pallor-Baseline | 1.8 (0.69) | 1.8 (0.70)
  Pallor-Change From Baseline to Week 12: number analyzed (Participants) | 212 | 217
  Pallor-Change From Baseline to Week 12 | -0.6 (0.75) | -0.9 (0.84)
  Pallor-Change From Baseline to Final Assessment: number analyzed (Participants) | 227 | 233
  Pallor-Change From Baseline to Final Assessment | -0.6 (0.75) | -0.9 (0.85)
  Dryness-Baseline | 1.8 (0.68) | 1.8 (0.75)
  Dryness-Change From Baseline to Week 12: number analyzed (Participants) | 212 | 217
  Dryness-Change From Baseline to Week 12 | -0.5 (0.85) | -0.9 (0.94)
  Dryness-Change From Baseline to Final Assessment: number analyzed (Participants) | 227 | 233
  Dryness-Change From Baseline to Final Assessment | -0.5 (0.83) | -0.9 (0.95)
  Friability-Baseline | 1.1 (0.93) | 1.2 (0.99)
  Friability-Change From Baseline to Week 12: number analyzed (Participants) | 212 | 217
  Friability-Change From Baseline to Week 12 | -0.6 (0.95) | -1.0 (0.99)
  Friability-Change From Baseline to Final Assessment: number analyzed (Participants) | 227 | 233
  Friability-Change From Baseline to Final Assessment | -0.6 (0.95) | -1.0 (0.97)
  Petechiae-Baseline | 0.7 (0.83) | 0.8 (0.89)
  Petechiae-Change From Baseline to Week 12: number analyzed (Participants) | 212 | 217
  Petechiae-Change From Baseline to Week 12 | -0.3 (0.78) | -0.6 (0.86)
  Petechiae-Change From Baseline to Final Assessment: number analyzed (Participants) | 227 | 233
  Petechiae-Change From Baseline to Final Assessment | -0.3 (0.78) | -0.6 (0.85)

9. Secondary Outcome: Change From Baseline in Vaginal pH to Week 12
Description: Vaginal pH was obtained at baseline and final visit of the study. The pH was a numeric value from 0 to 14 expressing the acidity or alkalinity of the vaginal fluids where 7 was neutral, lower values were more acidic (values of 0-6) and higher values more alkaline (values of 8-14). A negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
Number analyzed (Participants) | 233 | 239
score on a scale
  Baseline | 6.35 (0.66) | 6.37 (0.66)
  Change From Baseline to Week 12: number analyzed (Participants) | 211 | 216
  Change From Baseline to Week 12 | -0.53 (0.93) | -1.35 (0.89)

10. Secondary Outcome: Change From Baseline in the Percentage of Vaginal Superficial Cells to Week 12
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of superficial cells. A positive change from Baseline indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
Number analyzed (Participants) | 233 | 239
percentage of superficial cells
  Baseline | 0.2 (0.75) | 0.2 (0.70)
  Change From Baseline to Week 12: number analyzed (Participants) | 204 | 198
  Change From Baseline to Week 12 | 1.2 (5.35) | 10.5 (17.19)

11. Secondary Outcome: Change From Baseline in the Percentage of Vaginal Parabasal Cells to Week 12
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of parabasal cells. A negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
Number analyzed (Participants) | 233 | 239
percentage of parabasal cells
  Baseline | 50.6 (43.09) | 53.5 (42.00)
  Change From Baseline to Week 12: number analyzed (Participants) | 204 | 198
  Change From Baseline to Week 12 | -14.9 (39.88) | -48.2 (45.65)

ADVERSE EVENTS:
Time Frame: Up to Week 12
Description: Safety population included participants who were randomized into the study and took at least 1 dose of study drug.
Arm/Group | Vehicle (3 Times/Week) | WC3011 Estradiol Vaginal Cream (3 Times/Week)
All-Cause Mortality (participants affected / at risk) | 0/271 | 0/277
Serious Adverse Events (participants affected / at risk) | 1/271 | 3/277
Other Adverse Events (participants affected / at risk) | 42/271 | 38/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (3 Times/Week) (N=271) | WC3011 Estradiol Vaginal Cream (3 Times/Week) (N=277)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 1
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (3 Times/Week) (N=271) | WC3011 Estradiol Vaginal Cream (3 Times/Week) (N=277)
Urinary tract infection (Infections and infestations) | 21 | 10
Application site pain (General disorders) | 15 | 9
Vulvovaginal mycotic infection (Infections and infestations) | 9 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.